CLINICAL TRIAL: NCT04287985
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Efficacy and Safety of VIS649 in Participants With Immunoglobulin A (IgA) Nephropathy
Brief Title: Safety and Efficacy Study of VIS649 for IgA Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIS649-201; 2019-002531-29 (EudraCT Number); U1111-1263-1268 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2020-02-10; First posted 2020-02-27 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Immunoglobulin A Nephropathy; Glomerular Disease; IgAN
Keywords: VIS649; Kidney Diseases; Glomerulonephritis, IGA; Glomerulonephritis; Nephritis; Autoimmune Diseases; Immune System Diseases; Immunoglobulins; Antibodies; Immunoglobulin A; Immunologic Factors; Physiological Effects of Drugs; Proteinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases; Glomerulonephritis; Nephritis; Autoimmune Diseases; Immune System Diseases; Proteinuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, Investigator, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo, normal saline (0.9% NaCl) will be administered IV
  Interventions: Drug: Dose-Placebo
- Low Dose - VIS649 (Experimental): Low dose of VIS649 administered IV
  Interventions: Drug: Low Dose-VIS649
- Medium Dose - VIS649 (Experimental): Medium dose of VIS649 administered IV
  Interventions: Drug: Medium Dose-VIS649
- High Dose - VIS649 (Experimental): High dose of VIS649 administered IV
  Interventions: Drug: High Dose-VIS649

INTERVENTIONS:
Drug: Dose-Placebo — Unit Dose Strength - 0.9%.
  Arms: Placebo
Drug: Low Dose-VIS649 — Dose Level = Low
  Arms: Low Dose - VIS649
Drug: Medium Dose-VIS649 — Dose Level = Medium
  Arms: Medium Dose - VIS649
Drug: High Dose-VIS649 — Dose Level = High
  Arms: High Dose - VIS649

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VIS649 in participants with immunoglobulin A (IgA) Nephropathy (IgAN)

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, randomized, placebo-controlled study in patients aged 18 years and above with biopsy confirmed diagnosis of IgAN. The study is designed to test the safety and effectiveness of multiple doses of VIS649. The main objectives are to evaluate the safety and tolerability of VIS649 and to evaluate the dose response of different doses of VIS649 by measuring proteinuria.

The study is comprised of three main periods, Screening, Treatment (12 months) and Follow-Up (4 months). Approximately 144 patients will be enrolled. The findings from this study will form the basis for subsequent clinical development of VIS649.

VIS649 is a humanized immunoglobulin G (IgG2) monoclonal antibody that binds to and blocks the biological actions of the cytokine A PRoliferation Inducing Ligand (APRIL), a key factor in the production of aberrantly glycosylated IgA1 (a-g- IgA1), which is critical to the pathogenesis of IgAN.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participant is a male or female ≥ 18 years of age at the time of signing the informed consent.
2. Participant must have biopsy-confirmed IgAN.
3. Participant has medical records showing they have been on stable and maximally tolerated doses of either ACEI or ARB, as per local SOC and applicable guidelines, for at least 3 months preceding screening. Participants should optimally be on at least 50% of the maximum recommended dose of these agents; however, if a participant is on their maximally tolerated dose (and this is < 50% of the maximum recommended dose) and has been on this dose for at least 3 months, they may be enrolled. Participants who are unable to tolerate ACEI/ARB therapy may be eligible for participation in the study if their overall management of IgAN, including BP control, is as per local SOC and applicable guidelines.
4. Participants must have screening uPCR ≥ 0.75 g/g measured from a 24-hour urine or 24-hour urine protein ≥ 1.0 g/d, as measured from 24-hour urine collection. The proteinuria should be assessed when the participant is considered to be in a steady state with no recent heavy exercise, fever, or other potential issues that could impact the result.
5. Participants must have eGFR ≥ 45 mL/min/1.73 m² using the CKD-EPI formula.
6. Participant's serum Ig values must meet specified criteria
7. Female participants of childbearing potential must have a negative serum pregnancy test prior to the first dose.
8. Participant is willing to adhere to contraceptive requirements.
9. Participant or a legally authorized representative is able and is willing to give voluntary written informed consent

Exclusion Criteria:

Participants are excluded from the study if they meet any of the following criteria:

1. Participant has secondary forms of IgAN as defined by the treating physician.
2. Participant has co-existing CKD, other than IgAN.
3. Participant has evidence of additional pathological findings in the kidney biopsy (eg, diabetic kidney disease, membranous nephropathy, or lupus nephritis). However, hypertensive vascular changes are acceptable.
4. Participant has kidney biopsy MEST or MEST-C score as defined in the protocol.
5. Participant has nephrotic syndrome.
6. Participant has received a solid organ transplant, including kidney.
7. Participant has received bone marrow or hematologic stem cell transplantation.
8. Participant is currently receiving systemic immunosuppression (excluding topical, ophthalmic, per rectum, or inhaled corticosteroids).
9. Participant has received treatment with systemic corticosteroid therapy within 16 weeks of initial screening.
10. Participant has received treatment with a systemic immunosuppressive agents within 16 weeks of initial screening.
11. Participant has any chronic infectious disease.
12. Participant has acute infectious disease at the time of screening.
13. Participant has Type 1 diabetes.
14. Participant has uncontrolled Type 2 diabetes, as evidenced by a screening hemoglobin A1c value > 8%.
15. Participant has uncontrolled BP (> 140 mm Hg systolic or > 90 mm Hg diastolic)
16. Participant has a history of chronic autoimmune neurodegenerative disorder such as multiple sclerosis.
17. Participant has a known allergy or intolerance to any component of the study intervention.
18. Participant is breastfeeding.
19. Participant has poorly compensated or controlled ischemic heart disease or cardiomyopathy, as judged by the Investigator.
20. Participant has chronic obstructive pulmonary disease (COPD) or asthma that has required systemic steroid therapy during the prior year.
21. Participant has known cirrhosis or liver dysfunction, defined as presence of coagulopathy, platelet count < 100,000/μL or alanine aminotransferase > 3× upper limit of normal.
22. Participant has active malignancy or is receiving chemotherapy for malignancy, except for nonmelanoma skin cancers and cervical carcinoma in situ. Participants with prior malignancy who have been documented to be cancer-free for ≥ 5 years may be enrolled.
23. Participant is planning or scheduled to undergo a tonsillectomy. Prior tonsillectomy is acceptable (if greater than 6 months prior to screening).
24. Participant enrolled in another investigational drug or device study within 3 months prior to initial screening.
25. Participant with a pre-existing illness other than those listed above that, in the opinion of the Investigator, would place the participant at increased risk through participation in this study.
26. Participant is unable to comply with study protocol procedures and/or study visit schedules.
27. Participant with known or suspected alcohol or drug abuse that would compromise their safety or study participation of the participant, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asher Schachter, M.D., Study Director — Visterra, Inc.
Locations (83):
- United States (16):
  - Visterra Investigational Site, Birmingham, Alabama
  - Visterra Investigational Site, Los Angeles, California
  - Visterra Investigational Site, Oxnard, California
  - Visterra Investigational Site, Palo Alto, California
  - Visterra Investigational Site, Stanford, California
  - Visterra Investigational Site, Denver, Colorado
  - Visterra Investigational Site, Lawrenceville, Georgia
  - Visterra Investigational Site, Baton Rouge, Louisiana
  - Visterra Investigational Site, New Orleans, Louisiana
  - Visterra Investigational Site, Baltimore, Maryland
  - Visterra Investigational Site, Tupelo, Mississippi
  - Visterra Investigational Site, New York, New York
  - Visterra Investigational Site, Chapel Hill, North Carolina
  - Visterra Investigational Site, Columbus, Ohio
  - Visterra Investigational Site, Bethlehem, Pennsylvania
  - Visterra Investigational Site, Houston, Texas
- Australia (4):
  - Visterra Investigational Site, New Lambton Heights, New South Wales
  - Visterra Investigational Site, Saint Leonards, New South Wales
  - Visterra Investigational Site, Nambour, Queensland
  - Visterra Investigational Site, Nedlands, Western Australia
- Canada (3):
  - Visterra Investigational Site, Calgary, Alberta
  - Visterra Investigational Site, Brampton, Ontario
  - Visterra Investigational Site, Montreal, Quebec
- Hong Kong (4):
  - Visterra Investigational Site, Hong Kong, HK
  - Visterra Investigational Site, Hong Kong
  - Visterra Investigational Site, Kowloon
  - Visterra Investigational Site, Tsuen Wan
- India (10):
  - Visterra Investigational Site, Chandigarh, Chandigarh
  - Visterra Investigational Site, Bangalore, Karnataka
  - Visterra Investigational Site, Bengaluru, Karnataka
  - Visterra Investigational Site, Manipal, Karnataka
  - Visterra Investigational Site, Kozhikode, Kerala
  - Visterra Investigational Site, Thiruvananthapuram, Kerala
  - Visterra Investigational Site, New Delhi, National Capital Territory of Delhi
  - Visterra Investigational Site, Vellore, Tamil Nadu
  - Visterra Investigational Site, Hyderabad, Telangana
  - Visterra Investigational Site, Raebareli, Uttar Pradesh
- Japan (11):
  - Visterra Investigational Site, Toyoake-shi, Aichi-ken
  - Visterra Investigational Site, Tokyo, Nerima Ku
  - Visterra Investigational Site, Ashikaga, Tochigi
  - Visterra Investigational Site, Ashikaga-Shi
  - Visterra Investigational Site, Bunkyō City
  - Visterra Investigational Site, Kashihara-shi
  - Visterra Investigational Site, Minatoku
  - Visterra Investigational Site, Niigata
  - Visterra Investigational Site, Shinjuku-Ku
  - Visterra Investigational Site, Tsukuba
  - Visterra Investigational Site, Urayasu-Shi
- Malaysia (4):
  - Visterra Investigational Site, Klang
  - Visterra Investigational Site, Kuala Lumpur
  - Visterra Investigational Site, Kuantan
  - Visterra Investigational Site, Seremban
- Philippines (2):
  - Visterra Investigational Site, Diliman
  - Visterra Investigational Site, Quezon City
- Visterra Investigational Site, Singapore, Singapore
- South Korea (7):
  - Visterra Investigational Site, Seoul, Dongdaemun-gu
  - Visterra Investigational Site, Anyang-si, Gyeonggi-do
  - Visterra Investigational Site, Anyang
  - Visterra Investigational Site, Gangdong
  - Visterra Investigational Site, Hwaseong-si
  - Visterra Investigational Site, Seongnam-si
  - Visterra Investigational Site, Seoul
- Spain (8):
  - Visterra Investigational Site, L'Hospitalet de Llobregat, B
  - Visterra Investigational Site, Santander, CB
  - Visterra Investigational Site, Córdoba, CO
  - Visterra Investigational Site, Seville, SE
  - Visterra Investigational Site, Barcelona
  - Visterra Investigational Site, Madrid
  - Visterra Investigational Site, Seville
  - Visterra Investigational Site, Valencia
- Sri Lanka (3):
  - Visterra Investigational Site, Colombo
  - Visterra Investigational Site, Kandy
  - Visterra Investigational Site, Nugegoda
- Taiwan (4):
  - Visterra Investigational Site, Kaohsiung City
  - Visterra Investigational Site, Keelung
  - Visterra Investigational Site, New Taipei City
  - Visterra Investigational Site, Xitun
- Thailand (3):
  - Visterra Investigational Site, Bangkok
  - Visterra Investigational Site, Chiang Mai
  - Visterra Investigational Site, Ratchathewi
- United Kingdom (3):
  - Visterra Investigational Site, Bradford
  - Visterra Investigational Site, London
  - Visterra Investigational Site, Salford

REFERENCES:
- [Result] Mathur M, Barratt J, Chacko B, Chan TM, Kooienga L, Oh KH, Sahay M, Suzuki Y, Wong MG, Yarbrough J, Xia J, Pereira BJG; ENVISION Trial Investigators Group. A Phase 2 Trial of Sibeprenlimab in Patients with IgA Nephropathy. N Engl J Med. 2024 Jan 4;390(1):20-31. doi: 10.1056/NEJMoa2305635. Epub 2023 Nov 2. PMID 37916620
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639

RESULTS

PARTICIPANT FLOW:
Groups:
- VIS649 2 mg/kg: 2 mg/kg VIS649 administered intravenously
- VIS649 4 mg/kg: 4 mg/kg of VIS649 administered intravenously
- VIS649 8 mg/kg: 8 mg/kg of VIS649 administered intravenously
- Placebo: Placebo administered intravenously
Period: Overall Study
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Started | 38 | 41 | 38 | 38
Completed | 35 | 39 | 37 | 35
Not Completed | 3 | 2 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo | Total
Number analyzed (Participants) | 38 | 41 | 38 | 38 | 155
Age, Continuous [Median (Full Range); unit: Years] | 41.0 [25 to 71] | 39.0 [20 to 73] | 41.5 [23 to 72] | 36.5 [18 to 52] | 39.0 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 12 | 24 | 67
  Male | 22 | 26 | 26 | 14 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 2 | 9
  Not Hispanic or Latino | 36 | 38 | 35 | 35 | 144
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 28 | 31 | 28 | 28 | 115
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 9 | 9 | 8 | 10 | 36
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Japan | 5 | 5 | 5 | 4 | 19
  Australia | 1 | 2 | 0 | 3 | 6
  Canada | 0 | 1 | 1 | 0 | 2
  Hong Kong | 3 | 0 | 0 | 2 | 5
  India | 5 | 10 | 10 | 14 | 39
  South Korea | 2 | 4 | 5 | 4 | 15
  Malaysia | 3 | 2 | 2 | 1 | 8
  Philippines | 1 | 2 | 1 | 0 | 4
  Singapore | 1 | 3 | 2 | 0 | 6
  Spain | 2 | 3 | 1 | 3 | 9
  Sri Lanka | 2 | 1 | 1 | 1 | 5
  Taiwan | 0 | 0 | 1 | 0 | 1
  Thailand | 4 | 3 | 1 | 2 | 10
  United Kingdom | 1 | 0 | 2 | 2 | 5
  United States | 8 | 5 | 6 | 2 | 21
Height [Mean (Standard Deviation); unit: Centimeters] | 165.87 (8.919) | 167.50 (9.933) | 165.48 (10.277) | 161.84 (10.794) | 165.22 (10.120)
Weight [Mean (Standard Deviation); unit: Kilograms] | 74.97 (15.031) | 79.18 (21.216) | 75.54 (19.237) | 72.40 (21.124) | 75.59 (19.323)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.15 (4.529) | 28.10 (6.424) | 27.57 (5.778) | 27.35 (6.749) | 27.56 (5.894)
History of Hypertension [Count of Participants; unit: Participants] | 29 | 31 | 28 | 24 | 112
Time since biopsy [Median (Full Range); unit: Days] — Median. Count of days.
  Days | 781.0 [2 to 5657] | 288.0 [12 to 6263] | 364.0 [10 to 5776] | 933.0 [10 to 6431] | 565.0 [2 to 6431]
ACEI or ARB Therapy [Count of Participants; unit: Participants] — ACEI = angiotensin-converting enzyme inhibitor; ARB = angiotensin receptor blocker
  Participants | 37 | 40 | 37 | 38 | 152
SGLT2i use at baseline [Count of Participants; unit: Participants] — Participants taking sodium-glucose contransporter-2 inhibitor
  Participants | 3 | 2 | 1 | 3 | 9
Previous use of systemic immunosuppressive therapy [Count of Participants; unit: Participants] | 14 | 7 | 8 | 7 | 36
Baseline urinary protein excretion (mg/day) [Median (Full Range); unit: mg per day] | 1470.50 [668.0 to 6922.0] | 1927.00 [331.0 to 8600.0] | 1900.00 [764.0 to 12435.0] | 2133.50 [761.0 to 8479.0] | 1900 [331.0 to 12435.0]
Baseline 24-hour uPCR [Geometric Mean (Standard Deviation); unit: urinary protein/creatinine ratio] — uPCR = urinary protein/creatinine ratio
  urinary protein/creatinine ratio | 1.46 (0.123) | 1.53 (0.123) | 1.44 (0.137) | 1.68 (0.175) | 1.52 (0.069)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Graded by Severity
Description: The number of participants who experienced adverse events, graded by maximum severity, are presented.
Time Frame: Baseline to End of Study (16 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
Participants
  TEAE with a maximum severity of mild | 19 | 22 | 22 | 23
  TEAE with a maximum severity of moderate | 7 | 9 | 8 | 3
  TEAE with a maximum severity of severe | 2 | 2 | 1 | 1
  TEAE related to trial drug | 7 | 7 | 4 | 5
  TEAE related to trial drug with a maximum severity of Mild | 7 | 7 | 3 | 5
  TEAE related to trial drug with a maximum severity of Moderate | 0 | 0 | 1 | 0
  TEAE related to trial drug with a maximum severity of Severe | 0 | 0 | 0 | 0
  Serious TEAE | 2 | 2 | 1 | 2
  Serious TEAE related to trial drug | 0 | 0 | 0 | 0
  TEAE leading to trial drug interrupted | 5 | 1 | 3 | 0
  TEAE leading discontinuation of trial drug | 1 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 1

2. Primary Outcome: Changes From Baseline in Clinical Laboratory Tests
Description: The number of participants who experience a shift from normal at baseline to Grade 3/4 (moderate/sever) at a postbaseline time point are presented.
Time Frame: Baseline to End of Study (16 months)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
Participants
  Calcium | 1 | 0 | 0 | 0
  Potassium | 2 | 1 | 1 | 0
  Phosphate | 1 | 0 | 0 | 1
  Sodium | 0 | 1 | 0 | 0
  Triglycerides | 0 | 1 | 0 | 0
  Hemoglobin | 0 | 0 | 1 | 0

3. Primary Outcome: Clinically Meaningful Changes From Baseline in Vital Signs
Description: The number of participants who experienced clinically meaningful changes from baseline in vital signs (body mass index, diastolic blood pressure, height, heart rate, mean arterial pressure, respiratory rate, systolic blood pressure, temperature, and weight) are presented.
Time Frame: Baseline to End of Study (16 months)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 48
Participants | 0 | 0 | 0 | 2

4. Primary Outcome: Clinically Significant Physical Examinations
Description: Clinically significant physical examination findings are presented.
Time Frame: Baseline to End of Study (16 months)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
Participants | 1 | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in uPCR: Month 12
Description: Natural Log 24-Hour uPCR (Schedule A Urine Collection) Change from Baseline at Month 12: mixed model with repeated measurements
Time Frame: 12 months
Population: modified intent-to-treat (mITT) Population
Measure: Least Squares Mean (Standard Error); unit: g/g
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
g/g | -0.64 (0.2) | -0.89 (0.1) | -0.97 (0.2) | -0.22 (0.2)

6. Secondary Outcome: Change From Baseline in uPCR: Months 9 and 16
Description: Change from baseline in uPCR (Urine protein/creatinine ratio)
Time Frame: Baseline to 9 months and 16 months (16 months total)
Population: modified intent-to-treat (mITT) Population
Measure: Least Squares Mean (Standard Error); unit: g/g
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
g/g
  Month 9 | -0.70 (0.2) | -0.85 (0.1) | -0.99 (0.1) | -0.17 (0.2)
  Month 16 | -0.45 (0.2) | -0.87 (0.2) | -1.04 (0.2) | -0.11 (0.2)

7. Secondary Outcome: Change in 24-hour Urine Protein Excretion: Months 12 and 16
Description: Change in 24-hour urine protein excretion from baseline to Months 12 and 16
Time Frame: 16 months
Population: modified intent-to-treat (mITT) Population
Measure: Geometric Mean (95% Confidence Interval); unit: mg/day
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
mg/day
  Month 12 | 49.47 [30.6 to 63.2] | 57.80 [43.0 to 68.8] | 65.49 [53.1 to 74.6] | 18.74 [-11.5 to 40.8]
  Month 16 | 36.24 [10.7 to 54.5] | 55.19 [38.5 to 67.4] | 68.47 [56.3 to 77.2] | 8.30 [-28.1 to 34.4]

8. Secondary Outcome: Participants Achieving a Greater Than or Equal to 30% Decline From Baseline in uPCR at Months 9, 12, and 16
Description: Number of participants in each group achieving a greater than or equal to 30% decline from baseline in urinary protein/creatinine ratio (uPCR) at Months 9, 12, and 16
Time Frame: Baseline to 9,12, and 16 months (16 months total)
Population: modified intent-to-treat (mITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
Participants
  Month 9 | 19 | 20 | 21 | 7
  Month 12 | 19 | 24 | 23 | 11
  Month 16 | 18 | 21 | 24 | 8

9. Secondary Outcome: Participants in Each Group Achieving Clinical Remission
Description: Number of participants in each group achieving clinical remission. Clinical remission was defined as reduction in 24-hour urine protein excretion to less than 300 mg/day for at least 3 consecutive months.
Time Frame: Baseline to End of Study (16 months)
Population: modified intent-to-treat (mITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
Participants
  Month 9 | 4 | 5 | 7 | 1
  Month 12 | 3 | 5 | 10 | 1
  Month 16 | 3 | 7 | 9 | 1

10. Secondary Outcome: Change From Baseline in eGFR at Months 9, 12, and 16
Description: Change from baseline in (eGFR) at Months 9, 12, and 16
Time Frame: Baseline to 12 and 16 months
Population: modified intent-to-treat (mITT) Population
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
mL/min/1.73 m^2
  Month 12 (Day 360): number analyzed (Participants) | 34 | 39 | 36 | 38
  Month 12 (Day 360) | -2.35 (10.591) | 0.64 (9.212) | -1.25 (8.507) | -7.31 (14.318)
  Month 16 (Day 485): number analyzed (Participants) | 35 | 38 | 37 | 35
  Month 16 (Day 485) | -3.63 (10.132) | -0.18 (9.418) | -3.49 (9.503) | -8.54 (14.360)
  Month 9 (Day 270): number analyzed (Participants) | 35 | 41 | 37 | 36
  Month 9 (Day 270) | -0.26 (9.201) | 0.24 (7.519) | 0.16 (7.830) | -3.83 (14.062)

11. Secondary Outcome: Percent Change From Baseline in Total Serum IgA, IgG, and IgM Concentrations at Months 12 and 16
Description: Percent change from baseline in total serum immunoglobin (Ig)A, IgG, and IgM concentrations at Months 12 and 16 in PD population
Time Frame: Baseline to 12 and 16 months
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
Number analyzed (Participants) | 38 | 41 | 38 | 38
percentage change
  IgA : Month 12 (Day 360): number analyzed (Participants) | 34 | 37 | 35 | 36
  IgA : Month 12 (Day 360) | 48.35 (12.431) | 32.35 (10.403) | 31.07 (7.946) | 102.23 (10.584)
  IgA : Month 16 (Day 485): number analyzed (Participants) | 35 | 38 | 37 | 35
  IgA : Month 16 (Day 485) | 79.49 (12.167) | 69.62 (14.790) | 57.28 (14.645) | 101.22 (10.612)
  IgG : Month 12 (Day 360): number analyzed (Participants) | 34 | 38 | 35 | 36
  IgG : Month 12 (Day 360) | 72.88 (9.816) | 66.91 (12.613) | 65.40 (15.693) | 68.31 (13.218)
  IgG : Month 16 (Day 485): number analyzed (Participants) | 35 | 38 | 37 | 35
  IgG : Month 16 (Day 485) | 97.20 (10.006) | 96.00 (12.913) | 84.98 (20.144) | 101.48 (12.840)
  IgM : Month 12 (Day 360): number analyzed (Participants) | 34 | 38 | 35 | 36
  IgM : Month 12 (Day 360) | 37.33 (13.279) | 30.55 (11.959) | 30.03 (8.017) | 98.21 (13.656)
  IgM : Month 16 (Day 485): number analyzed (Participants) | 35 | 38 | 37 | 35
  IgM : Month 16 (Day 485) | 85.67 (10.729) | 84.74 (20.481) | 62.51 (16.864) | 97.45 (13.239)

12. Secondary Outcome: Mean Serum PK Parameters at Month 0 and Month 11: Cmax
Description: Serum PK parameters: maximum serum concentration (Cmax)
Time Frame: Months 0 and 11
Population: Intensive Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg
Number analyzed (Participants) | 38 | 41 | 38
μg/mL
  Month 0: number analyzed (Participants) | 6 | 10 | 8
  Month 0 | 78.78 (16.69) | 128.88 (38.52) | 245.75 (46.35)
  Month 11: number analyzed (Participants) | 4 | 8 | 8
  Month 11 | 65.45 (21.83) | 185.63 (54.29) | 939.13 (1140.10)

13. Secondary Outcome: Median Serum PK Parameters at Month 0 and Month 11: Tmax
Description: Serum PK parameters: time of maximum serum concentration (Tmax)
Time Frame: Month 0 and Month 11
Population: Intensive Pharmacokinetic Population
Measure: Median (Full Range); unit: days
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg
Number analyzed (Participants) | 38 | 41 | 38
days
  Tmax: Month 0: number analyzed (Participants) | 6 | 10 | 8
  Tmax: Month 0 | 0.052 [0.05 to 0.14] | 0.052 [0.04 to 0.13] | 0.125 [0.05 to 0.13]
  Tmax: Month 11: number analyzed (Participants) | 4 | 8 | 8
  Tmax: Month 11 | 0.089 [0.05 to 0.13] | 0.127 [0.05 to 8.00] | 0.123 [0.05 to 19.99]

14. Secondary Outcome: Mean Serum PK Parameters at Month 0: AUC0-inf and AUC0-30
Description: Serum PK parameters of area under the concentration-time curve from time 0 to infinity (AUC0-inf) and area under the concentration-time curve from time 0 to Day 30 (AUC0-30)
Time Frame: Month 0
Population: Intensive pharmacokinetic population
Measure: Mean (Standard Deviation); unit: day∙μg/mL
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg
Number analyzed (Participants) | 38 | 41 | 38
day∙μg/mL
  AUC0-inf: number analyzed (Participants) | 5 | 6 | 0
  AUC0-inf | 544.49 (191.80) | 1189.68 (184.72) |
  AUC0-30: number analyzed (Participants) | 6 | 10 | 8
  AUC0-30 | 542.69 (167.88) | 1245.02 (311.85) | 3019.78 (473.59)

15. Secondary Outcome: Mean Serum PK Parameters at Month 0 and Month 11: t1/2z
Description: Serum PK parameters: terminal elimination half-life(t1/2z)
Time Frame: Month 0 and Month 11
Population: Intensive Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg
Number analyzed (Participants) | 38 | 41 | 38
days
  Month 0: number analyzed (Participants) | 6 | 9 | 7
  Month 0 | 5.78 (1.25) | 10.87 (3.23) | 18.64 (5.26)
  Month 11: number analyzed (Participants) | 2 | 7 | 7
  Month 11 | 8.82 (2.89) | 10.67 (2.66) | 14.85 (8.32)

16. Secondary Outcome: Median Serum PK Parameters at Month 0: CL
Description: Serum PK parameters of clearance.
  8 mg/kg was not reported for this outcome measure. Other arms were not provided due to participants meeting exclusion criteria: %AUCext > 20% and R2 Adjusted < 0.8. Affected parameters at participant visits meeting this criteria were excluded.
Time Frame: Month 0
Population: Intensive pharmacokinetic population
Measure: Median (Standard Deviation); unit: mL/day
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg
Number analyzed (Participants) | 5 | 6
mL/day | 257.89 (71.77) | 315.94 (95.36)

17. Secondary Outcome: Mean Serum PK Parameters at Month 0: Vz
Description: Serum PK parameters of apparent volume of distribution (Vz).
  8 mg/kg was not reported for this outcome measure. Other arms were not provided due to participants meeting exclusion criteria: %AUCext > 20% and R2 Adjusted < 0.8. Affected parameters at participant visits meeting this criteria were excluded.
Time Frame: Month 0
Population: Intensive pharmacokinetic population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg
Number analyzed (Participants) | 5 | 6
mL | 2056.05 (726.38) | 4075.62 (1184.26)

18. Secondary Outcome: Mean Serum PK Parameters at Month 11: AUCτ
Description: Serum PK parameters: area under the concentration-time curve from time 0 to the end of the dosing period (AUCτ)
Time Frame: Month 11
Population: Intensive Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: day∙μg/mL
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg
Number analyzed (Participants) | 3 | 8 | 8
day∙μg/mL | 555.17 (116.13) | 2403.14 (929.12) | 13057.23 (8432.07)

19. Secondary Outcome: Mean Serum PK Parameters at Month 11: Vss
Description: Serum PK parameters: volume of distribution at steady-state (Vss)
Time Frame: Month 11
Population: Intensive Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg
Number analyzed (Participants) | 2 | 7 | 7
mL/kg | 2998.81 (1437.79) | 2670.87 (854.09) | 2517.15 (1529.85)

20. Secondary Outcome: Mean Serum PK Parameters at Month 11: CLss
Description: Serum PK parameters: clearance at steady-state (CLss)
Time Frame: Month 11
Population: Intensive Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg
Number analyzed (Participants) | 3 | 8 | 8
mL/day | 227.66 (50.99) | 176.22 (69.07) | 60.55 (25.82)

21. Secondary Outcome: Mean Serum PK Parameters at Month 11: Rac[AUC0-30]
Description: Serum PK parameters: accumulation ratio of area under the concentration-time curve from time 0 to infinity (Rac[AUC0-30])
Time Frame: Month 11
Population: Intensive Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg
Number analyzed (Participants) | 3 | 8 | 8
ratio | 1.27 (0.02) | 2.01 (0.63) | 4.41 (3.08)

ADVERSE EVENTS:
Time Frame: Baseline to End of Study (16 months).
Description: Adverse events were collected from screening through the M16 (or EOS) visit, up to 485 days. Collection methods were both systematic (at clinical visits) and non-systematic (reported by the patient). The protocol used standard terminology for determining adverse events and serious adverse events. The intensity of the events was assessed by the Investigator as either "mild," "moderate," or "severe."
Arm/Group | VIS649 2 mg/kg | VIS649 4 mg/kg | VIS649 8 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41 | 0/38 | 1/38
Serious Adverse Events (participants affected / at risk) | 2/38 | 2/41 | 1/38 | 2/38
Other Adverse Events (participants affected / at risk) | 28/38 | 33/41 | 31/38 | 27/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIS649 2 mg/kg (N=38) | VIS649 4 mg/kg (N=41) | VIS649 8 mg/kg (N=38) | Placebo (N=38)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Henoch-Schonlein tissue disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIS649 2 mg/kg (N=38) | VIS649 4 mg/kg (N=41) | VIS649 8 mg/kg (N=38) | Placebo (N=38)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 0
Cataract nuclear (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Episcleritis (Eye disorders) | 0 | 1 | 0 | 0
Eyelids pruritus (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 2 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0
Induration (General disorders) | 1 | 0 | 0 | 0
Infusion site discomfort (General disorders) | 0 | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 0 | 1
Infusion site thrombosis (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 1
Oedema peripheral (General disorders) | 4 | 1 | 0 | 1
Pain (General disorders) | 2 | 0 | 2 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1
Puncture site pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 5 | 6 | 6
Swelling face (General disorders) | 0 | 0 | 1 | 1
Vaccination site discomfort (General disorders) | 0 | 1 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Dust allergy (Immune system disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 10 | 11 | 13 | 16
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1
Helminthic infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 5 | 6 | 3
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Systemic viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Human bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post vaccination fever (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Antithrombin III decreased (Investigations) | 1 | 0 | 0 | 0
Blood bicarbonate abnormal (Investigations) | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 2 | 0 | 1
Coronavirus test positive (Investigations) | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 3 | 0
Vitamin D decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Asterixis (Nervous system disorders) | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 1 | 2
Headache (Nervous system disorders) | 1 | 5 | 3 | 4
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 1
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 3 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements are in place that restrict investigators from publishing the results of the trial.

DOCUMENTS (4):
  • Study Protocol: Version 4 (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04287985/Prot_000.pdf
  • Study Protocol: Version 3 (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT04287985/Prot_001.pdf
  • Study Protocol: Version 2 (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04287985/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT04287985/SAP_003.pdf